CLINICAL TRIAL: NCT05917054
Title: Comparison of Bipolar Vascular Sealing and Conventional Back-table Dissection in Terms of Post-renal Transplant Drainage and Back-table Preparation Times
Brief Title: Comparison of Bipolar Vascular Sealing and Conventional Back-table Dissection
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Other Study IDs: 2/2021.K-66
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Drain Site Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1-bipolar sealing: During the back-table preparation stage of these kidney transplant recipients, bipolar sealing method will be used for sealing the small vessels and lymphatics of the renal allograft.
  Interventions: Other: use of bipolar vascular sealing method on the renal allograft at the back-table stage
- Group 2-conventional silk tie: During the back-table preparation stage of these kidney transplant recipients, conventional silk-tie method will be used for sealing the small vessels and lymphatics of the renal allograft.
  Interventions: Other: use of bipolar vascular sealing method on the renal allograft at the back-table stage

INTERVENTIONS:
Other: use of bipolar vascular sealing method on the renal allograft at the back-table stage — Ligation of small vessels and lymphatics of the renal graft at the back-table stage prior to transplantation to the recipient is a routine practice in kidney transplantation. Bipolar vascular sealing method will be used for this purpose in Group 1, while the conventional silk-tie method will be used in Group 2.

SUMMARY:
The usage of vessel sealing devices has been gaining popularity in all surgical specialties. Post-renal transplant drain placement is a common practice among transplant surgeons. However, prolonged drainage accompanied by surgical wound complications and perirenal fluid collections is a frequent complication experienced by the recipients. This study aimed to compare bipolar sealing with conventional back-table dissection in terms of post-renal transplant drainage duration, amount, surgical wound complication, and back-table preparation time.

DETAILED DESCRIPTION:
Consecutive recipients receiving a living donor kidney transplant at Istinye University Organ Transplantation Center will be enrolled in this study. Istinye University Hospital Ethical Review Committee approved the clinical study (2/2021.K-66). Informed consent will be obtained from all individual participants included in this study. The recipients will be randomized into two groups by a simple randomization (i.e., flipping coin) method. In Group 1, bipolar sealing method will be used, and in Group 2, conventional silk tie ligature will be used during the back-table dissections of the harvested grafts. Data parameters including recipient age, gender, body mass index (BMI), cause of end-stage renal disease, dialysis modality, postoperative pain, surgical drainage duration, back-table time, cold ischemia time, and surgical site infections will be collected on a database by a research nurse. The exclusion criteria will be pediatric recipients and recipients who had received a kidney transplant previously. The donor nephrectomies will be performed using a pure laparoscopic technique. A standard right/left lower Gibson incision will be made in every recipient, and the renal bed will be prepared extraperitoneally. The external iliac vein and external iliac artery will be used for graft vessel anastomosis. Lymphatic vessels will be tied by 3/0 and 2/0 silk sutures in the conventional group, whereas bipolar sealing method will be used in the other.

Study investigators will be blinded to patient randomizations. All vascular anastomoses and bladder-ureter anastomoses will be performed by the primary surgeon (E.E). One closed-suction Hemovac drain will be placed at the lower pole of the graft in all recipients, and it will be removed when discharge is less than 50 ml over 24 hours. The Gregoir-Lich anti-reflux anastomosis technique performed all ureteroneocystostomies with Polydioxanone (PDS) sutures. A double J stent will be inserted in all cases. A Foley catheter will also be placed in the bladder and removed on the fourth postoperative day as recommended in the literature. All patients will be evaluated for pain on the postoperative 1 st day. The pain will be assessed with a visual analog scale, scoring from 0 to 10, with 0 being no pain and 10 being the worst pain ever experienced. Triple immunosuppression with tacrolimus, mycophenolate mofetil, and steroid will be initiated on post-renal transplant day 1 to all recipients. In addition, high-risk recipients will receive thymoglobulin as induction, while low-risk recipients will receive Basiliximab on days 0 and 4 post-transplant. All recipients will be anticoagulated by daily subcutaneous enoxaparin 0,6 cc injections starting on the day of surgery until the day of discharge. Patients will be followed in terms of pain, drainage length, and wound complications for 6 months. Surgical wounds will be assessed daily during the post-transplant 1 st week, then weekly afterward.

ELIGIBILITY:
Inclusion Criteria:

Adult (aged 18 or higher) patients who will undergo a live-donor kidney transplant surgery in Istinye University Hospital and consent to participation in this study.

Exclusion Criteria:

* Pediatric (age lower than 18) recipients
* Patients who received kidney transplant before

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult (aged 18 or higher) patients with end-stage renal disease scheduled for a live donor kidney transplantation and consent to participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Drainage duration | days
  Time between renal transplantation and removal of the surgical drain

SECONDARY OUTCOMES:
Wound complications | months
  Emergence of wound complications

CONTACTS AND LOCATIONS:
Overall Officials: Eryigit Eren, MD, Principal Investigator — Istinye University Training and Research Hospital
Locations (1):
- Istinye University Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No